CLINICAL TRIAL: NCT01721980
Title: Double-blind, Randomized, Placebo-controlled Study for the Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of GLPG0974 in Healthy Male Subjects
Brief Title: Multiple Ascending Dose Study of GLPG0974 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0974-CL-102
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
MeSH Terms: interventions — 4-(((R)-1-(benzo(b)thiophene-3-carbonyl)-2-methyl-azetidine-2-carbonyl)-(3-chloro-benzyl)-amino)-butyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50 mg GLPG0974 or placebo (Other): 50 mg GLPG0974 dose as oral capsule or placebo capsule, daily for 14 days
  Interventions: Drug: GLPG0974; Drug: Placebo
- 100 mg GLPG0974 or placebo (Other): 100 mg GLPG0974 dose as oral capsule or placebo oral capsule, daily for 14 days
  Interventions: Drug: GLPG0974; Drug: Placebo
- 200 mg GLPG0974 or placebo (Other): 200 mg GLPG0974 dose as oral capsule or placebo capsule, daily for 14 days
  Interventions: Drug: GLPG0974; Drug: Placebo
- 400 mg GLPG0974 or placebo (Other): 400 mg GLPG0974 dose as oral capsule or placebo capsule, daily for 14 days
  Interventions: Drug: GLPG0974; Drug: Placebo

INTERVENTIONS:
Drug: GLPG0974
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability after multiple ascending oral doses of GLPG0974 given to healthy male subjects for 14 days, compared to placebo.

Furthermore, during the course of the study, the amount of GLPG0974 present in the blood and urine (pharmacokinetics) as well as the effects of GLPG0974 on mechanism of action-related parameters in the blood and stool samples (pharmacodynamics) will be characterized compared to placebo.

Also, the effect of the compound on glucose tolerance will be explored as well as the potential of cytochrome P450 (CYP)3A4 induction by repeated dosing with GLPG0974.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG0974 in comparison with placebo after a single oral dose in healthy subjects in terms of adverse events, physical examinations, vital signs, ECG and lab assessments

SECONDARY OUTCOMES:
The amount of GLPG0974 in plasma and urine over time after multiple oral dose | Between Day 1 predose and Day 14
  To characterize the amount of GLPG0974 in plasma and urine over time - pharmacokinetics (PK) - after multiple oral doses in healthy subjects
Inhibition of CD11b on neutrophils in blood after multiple oral doses of GLPG0974 | Day 1 and Day 13, predose until 24h post dose
  To characterize the pharmacodynamics (PD) of GLPG0974 by means of inhibition of expression of CD11b on neutrophils after multiple oral doses in healthy subjects

OTHER OUTCOMES:
Ratio of 6b-hydroxycortisol/cortisol in urine | Predose and postdose on Day 1 and Day 13 for 24h
  Potential of CYP3A4 induction by repeated dosing with GLPG0974 will be assessed by means of the ratio of 6b-hydroxycortisol/cortisol in urine
Levels of faecal calprotectin in stool | Prior to first dosing and postdose (between Day 12 and 15)
  Concentrations of faecal calprotectin will be measured as a pharmacodynamic marker in a single stool sample predose and postdose
Glucose and insulin concentrations after glucose loading | Day -1 (predose) and Day 14 (postdose)
  Oral glucose tolerance test by means of measuring concentrations of glucose and insulin after glucose loading, once predosing and once postdosing of GLPG0974

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium